CLINICAL TRIAL: NCT06459440
Title: Effect of Group-Task-Oriented Training on Gross Motor and Fine Motor Functions and Activities of Daily Living Skills in Children With Downs Syndrome.
Brief Title: Effect of Group-Task-Oriented Training on GMFM and ADL in Children With DS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0791
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Downs Syndrome
Keywords: Down Syndrome, Group-Oriented task training, Motor skills
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: It will be randomized control trial in which non probability convenient sampling will be used. Two groups of 4-8 age will be formed in which participants will be randomly divided.Group A will be receive Group-Task-Oriented Training. Group B will be receive routine therapy.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Task Oriented Training (Experimental): All session will be give 4 days a week
  1.Week 1-2: Warm-up (10 mins) Core strengthening (10 mins) Posture training (10 mins) Balance training (10 mins)
  Week 3-4:
  Gross motor skills (10 mins) Fine motor skills (10 mins) Gait training (10 mins)
  Proprioception training (10 mins) Week 5-6 Activities of daily living (10 mins)
  Interventions: Behavioral: Group Task oriented Training
- Routine Treatment (Active Comparator): 1.Week 1-2 : Foundation building (4 sessions per week) Gentle stretching exercises (20 minutes). Basic strengthening exercises (20 minutes) (26). Weeks 3-4: Balance and coordination (4 sessions per week ) Balance exercises and core stability (20 minutes). Coordination drills (20 minutes) (26). Weeks 5-6: Functional activities (4 sessions per week )
  Incorporate functional activities into therapy (e.g., walking, reaching) (20 minutes) (26).
  Interventions: Other: Routine Treatment

INTERVENTIONS:
Behavioral: Group Task oriented Training — Group Task-Oriented Training for individuals with Down syndrome is an approach that focuses on improving specific skills and promoting social interaction through collaborative activities. This training method involves organizing individuals with Down syndrome into small groups to work on tasks that target various developmental areas, such as motor skills, communication, and socialization. The tasks are designed to be meaningful, engaging, and relevant to the participants' daily lives.
  Arms: Group Task Oriented Training
Other: Routine Treatment — 1.Week 1-2 : Foundation building (4 sessions per week) Gentle stretching exercises (20 minutes). Basic strengthening exercises (20 minutes) (26). Weeks 3-4: Balance and coordination (4 sessions per week ) Balance exercises and core stability (20 minutes). Coordination drills (20 minutes) (26). Weeks 5-6: Functional activities (4 sessions per week )
  Incorporate functional activities into therapy (e.g., walking, reaching) (20 minutes)
  Arms: Routine Treatment

SUMMARY:
Down syndrome, a genetic condition resulting from an additional copy of chromosome 21, manifests with distinct facial features and intellectual challenges. Individuals with Down syndrome often face delays in motor skills, speech, and language development, alongside potential health issues. Down syndrome commonly encounter difficulties in both gross and fine motor functions due to factors like low muscle tone. Nonetheless, targeted interventions, including physical, significantly enhance motor skills. Daily living activities for individuals with Down syndrome cover personal care and household tasks, with structured routines and consistent support fostering independence. Group Task-Oriented Training, focusing on skill improvement and social interaction through collaborative activities, offers a meaningful approach to enhancing the overall quality of life for individuals with Down syndrome.

DETAILED DESCRIPTION:
Group A receive Group-Task-Oriented Training. Group B receive routine therapy. Both the groups receive intervention for 40 minutes per session 4 times a week for six weeks.This study will be a randomized controlled trial and will be completed over a 10-month period in Lahore. Data will be collected from PSRD Hospital and Rising Sun Institute for Special Children. The estimated sample size is 44 participants, will be divided into two groups using non-probability convenient sampling. Inclusion criteria for Down syndrome children aged 4-8 include willingness to engage in Group-Task-Oriented Training sessions and stable health conditions. Exclusion criteria involve recent surgeries or severe medical conditions hindering participation. Data collection tools comprise the Jebsen hand function test, Gross Motor Function Measure, and Pediatric Evaluation of Disability Inventory.Participants are randomly assigned to an Experimental Group undergoing group task-oriented training and a Control Group receiving routine physical therapy. The training sessions for both groups are detailed, focusing on motor skills, fine motor function, gait training, and activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome children age ranged between 4-8 years (20).
* Both male and female genders are included (21).
* Children and their families willing to engage in Group-Task-Oriented Training sessions (20).
* Participants in stable health conditions suitable for engaging in the prescribed training program (20).

Exclusion Criteria:

* Any recent surgical procedure (21).
* Children with severe medical conditions or comorbidities that may interfere with participation in the Group-Task-Oriented Training (21).
* Children with severe physical limitations that could hinder active participation in the training sessions (21)

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
GROSS MOTOR FUNCTION MEASURE | 6 weeks
  The Gross Motor Function Measure (GMFM) is a clinical tool used to assess gross motor function in individuals with cerebral palsy. It evaluates five dimensions: lying and rolling, sitting, crawling and kneeling, standing, and walking, running, and jumping. Each dimension has specific items reflecting developmental motor milestones. Scoring is based on observed abilities, ranging from 0 (no ability) to 3 (complete ability). The total score indicates the individual's overall gross motor function. The GMFM is valuable for tracking progress over time and guiding intervention strategies for those with cerebral palsy (23).
Jebsen Hand function test | 6 weeks
  The Jebsen Hand Function Test (JHFT) is a clinical tool assessing hand function and fine motor skills in daily activities. Tasks include writing, card manipulation, and object handling. Widely used in rehabilitation, it measures speed and efficiency in completing tasks, aiding treatment planning for conditions affecting hand function. The JHFT demonstrates good reliability and validity, ensuring consistent and accurate assessment results, making it valuable for tracking progress and guiding interventions in individuals with upper extremity conditions
Pediatric Evaluation of Disability Inventory (PEDI) | 6 weeks
  The PEDI comprises three domains: self-care, mobility, and social function. Each domain evaluates specific tasks including feeding, dressing, walking, and communicating with others. It takes into consideration the child's age, developmental stage, and specific diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Sameen Fatima, MS*, Principal Investigator — Riphah International Univerisity
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Antonarakis SE, Skotko BG, Rafii MS, Strydom A, Pape SE, Bianchi DW, Sherman SL, Reeves RH. Down syndrome. Nat Rev Dis Primers. 2020 Feb 6;6(1):9. doi: 10.1038/s41572-019-0143-7. PMID 32029743